CLINICAL TRIAL: NCT03323281
Title: Impact of Cognitive, Psychological and Psychiatric Factors in Pathogenesis of Diabetic Foot and Recurrence : Study in Diabetic Patients
Brief Title: Neuropsychiatric Factors
Acronym: Diapepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: UF9805
Record Dates: First submitted 2017-05-16; First posted 2017-10-26 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
Keywords: Diabetic foot; Cognitive functions; Psychiatric disorders; Neurology; Psychiatry
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Type 1 or Type 2 with foot wound: Type 1 or type 2 diabetic patients with hospitalization for foot wounds having an interview with a neuropsychologist or a physician trained in neuropsychological assessments
  Interventions: Other: Neuropsychological assessments
- Diabetic Type 1 or Type 2 without a foot wound or antecedent: Type 1 or Type 2 diabetic patients with no foot wounds or history of foot wounds having an interview with a neuropsychologist or a physician trained in neuropsychological assessments
  Interventions: Other: Neuropsychological assessments

INTERVENTIONS:
Other: Neuropsychological assessments — Maintenance of approximately 1h30 with a neuropsychologist or a physician trained in neuropsychological assessments in Diabetic Type 1 or Type 2 with foot wound hospitalization and Diabetic Type 1 or Type 2 without a foot wound or antecedent Of foot wound (podological risk grade 0 to 2, including foot of Charcot)

SUMMARY:
It is estimated that approximately 20-25% of diabetic patients will have at least one trophic disorder during their period. The appearance of a trophic disorder in a diabetic patient is a serious complication, indicating that diabetes is often complicated. The consequences are serious for the patient with an impairment of his quality of life, but also for society with a high cost in terms of health care costs.

It should also be noted that diabetes remains the main cause of non-traumatic amputation in most developed countries, with amputation often preceded by a trophic disorder. In addition, 20% of amputees are re-amputated at least once a year. Thus, the consequences of diabetic foot injuries are important in human, social and health terms and are the subject of increased health care spending.

Many studies have shown that diabetes is a risk factor for dementia, whether it is Alzheimer's disease, Alzheimer's disease or the vascular component or pure vascular dementia.

However, an understanding of the cognitive mechanisms involved in the management of diabetes and in particular in the diabetic foot and its recurrence remains partial and no study has integrated the severity of the risk of the foot (evaluated by the podological risk) Specific implication of some Cognitive abilities, especially in relation to episodic memory, and social cognition integrating decision-making abilities. These specific disorders could have a major impact in diabetes follow-up, therapeutic adherence and the risk of developing recurrent trophic disorders.

Thus, the coexistence of diabetes with a mental pathology makes the management of the subject more complex and exposes it to more complications.

In the management of chronic diabetic disease, adherence to treatment is essential. It is therefore important to detect the specific effects of this type of personality on the prognosis of diabetes and the appearance of foot wounds.

DETAILED DESCRIPTION:
It is estimated that approximately 20-25% of diabetic patients will have at least one trophic disorder during their. The occurrence of a trophic disorder in a diabetic patient is a serious complication, indicating a diabetes often complicated. The consequences are severe for the patient with an alteration of his quality of life, but also for society with a high cost in terms of healthcare costs.

It should also be pointed out that diabetes is still the leading cause of non-traumatic amputation in most developped countries, with amputation often preceded by a trophic disorder. Further, 20% of amputees are re-amputed at least once a year. Thus the consequences of the wounds of the diabetic foot are important on the human, social and health level and are the subject of an increase of the health expenses.

Many studies have shown that diabetes is a risk factor for dementia whether it is Alzheimer's disease, Alzheimer's disease with vascular component or pure vascular dementia.

However, an understanding of the cognitive mechanisms involved in the management of diabetes and in particular in the diabetic foot and its recurrence remains partial and no study has integrated the severity of the foot risk (evaluated by the podological risk ) and the specific involvement of certain cognitive abilities, in particular in relation to episodic memory, and social cognition integrating decision-making abilities. These specific disorders could have a major implication in the follow-up of diabetes, in the therapeutic adherence and in the risk of developing recurrent trophic disorders.

Thus, the coexistence of diabetes with a mental pathology makes the management of the subject more complex and exposes it to more complications.

In the management of chronic diabetic disease, adherence to treatment is essential. It is therefore important to detect the specific effects of this type of personality on the prognosis of diabetes and the occurrence of foot wounds.

ELIGIBILITY:
Inclusion Criteria:

"Diabetic subjects with foot wounds"

* Subjects over 45 years old
* Diabetic type 1 or type 2 with foot wound (podological risk grade 3) in hospitalization in the Nutrition-Diabetes Unit CHU Lapeyronie or in the Department of Metabolic Diseases CHRU Grau du Roi.
* Having given their informed consent for the study

"Diabetic subjects without a foot wound"

* Subjects over 45 years old
* Type 1 or type 2 diabetics without a foot wound or previous foot wound (grade 0 to 2 grade, including Charcot foot) hospitalized or seen for consultation in the Nutrition-Diabetes Unit LaUyronie CHU or Metabolic Diseases CHRU Grau of the King.
* Having given their informed consent for the study

Exclusion Criteria:

* Patients who can not complete the self-questionnaires or can not carry out the cognitive tests (blindness, non-French speaking patient, illiteracy)
* Major physical or neurosensory problems that may interfere with the tests

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 133 diabetic subjects with foot wounds and 133 diabetic subjects without foot wounds
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2024-12-07 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Measuring memory | 1 day
  The test of Rappel libre/Rappel indicé à 16 items (RL/RI 16) : memory measure
  * Range : min :0 max:16
  * better or worse outcome according the population studied (age, education) (no cut off scores)

SECONDARY OUTCOMES:
Measuring memory | 2 years after the hospitalization
  The test of Rappel libre/Rappel indicé à 16 items (RL/RI 16) : memory measure
  * Range : min :0 max:16
  * better or worse outcome according the population studied (age, education) (no cut off scores)

OTHER OUTCOMES:
Measurement of cognition by the Mini Mental State Examination (MMSE) | 1 day
  Measures of cognition by the realization of Mini Mental State Examination (MMSE)
  * Range min :0 max 30
  * Score < or = 24 : cognitive disorders This test will be performed over 1 day during hospitalization
Weschler Cognition Measures | 1 day
  Weschler Cognition Measurements This test will be performed over 1 day during hospitalization
Measurement of cognition by the EMPAN direct and indirect | 1 day
  Measurement of cognition by the EMPAN direct and indirect EMPAN direct : Range : 1-8 and no cut off score EMPAN indirect : Range : 1-8 and no cut off score
  This test will be performed over 1 day during hospitalization
Measurement of cognition by the Trail Making A (TMTA) and Trail Making B (TMTB) | 1 day
  Measurement of cognition by the TMTA and TMTB Trail Making A : Range : 0-26 and no cut off score Trail Making B : Range : 0-13 and no cut off score This test will be performed over 1 day during hospitalization
Measurement of cognition by the phonemic verbal fluence | 1 day
  Measurement of cognition by the phonemic verbal fluence This test will be performed over 1 day during hospitalization
Measurement of cognition by the semantic verbal fluence | 1 day
  Measurement of cognition by the semantic verbal fluence This test will be performed over 1 day during hospitalization
Measurement of cognition by the phonemic verbal fluence | 2 years after the hospitalization
  Measurement of cognition by the phonemic verbal fluence
Measurement of cognition by the semantic verbal fluence | 2 years after the hospitalization
  Measurement of cognition by the semantic verbal fluence
Measurement of cognition by the the Trail Making A (TMTA) and Trail Making B (TMTB) | 2 years after the hospitalization
  Measurement of cognition by the TMTA and TMTB
  Trail Making A : Range : 0-26 and no cut off score Trail Making B : Range : 0-13 and no cut off score
Measurement of cognition by the empan direct and indirect | 2 years after the hospitalization
  Measurement of cognition by the EMPAN direct and indirect EMPAN direct : Range : 1-8 and no cut off score EMPAN indirect : Range : 1-8 and no cut off score
Weschler Cognition Measures | 2 years after the hospitalization
  Weschler Cognition Measurements
Measurement of cognition by the Mini Mental State Examination (MMSE) | 2 years after the hospitalization
  Measures of cognition by the realization of Mini Mental State Examination (MMSE)
  * Range min :0 max 30
  * Score < or = 24 : cognitive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC